CLINICAL TRIAL: NCT03494686
Title: Large Loop Excision of the Transformatione Zone Under General Versus Local Anesthesia: a Randomized Trial.
Brief Title: LLETZ Under General Versus Local Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zydolab - Institute of Cytology and Immune Cytochemistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONE-4
Record Dates: First submitted 2018-04-03; First posted 2018-04-11 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Uterine Cervical Dysplasia
Keywords: conization; LLETZ; randomized controlled trial; loop excision; general anaesthesia; local anaesthesia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLETZ under local anaesthesia (Experimental): The LLETZ procedure will be performed under local anaesthesia
  Interventions: Procedure: LLETZ under local anaesthesia
- LLETZ under general anaesthesia (Active Comparator): The LLETZ procedure will be performed under general anaesthesia
  Interventions: Procedure: LLETZ under general anaesthesia

INTERVENTIONS:
Procedure: LLETZ under local anaesthesia — Conization will be performed under local anaesthesia
  Arms: LLETZ under local anaesthesia
Procedure: LLETZ under general anaesthesia — Conization will be performed under general anaesthesia
  Arms: LLETZ under general anaesthesia

SUMMARY:
The investigators conduct a prospective, randomized trial to assess the benefits of performing large loop excision of the transformatione zone (LLETZ) under local anesthesia and compare it to LLETZ under general anesthesia. The primary endpoint of this study is women´s satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* colposcopy Prior to conization
* informed consent
* histologically proven high grade cervical dysplasia
* Transformation zone typ 1 or 2

Exclusion Criteria:

* significant language barrier
* a personal history of conization
* pregnancy
* the use of blood thinner
* unwillingness to participate
* oncological disease
* inpatient treatment
* women who are not fasting
* risk of aspiration
* columnar-squamous epithelium border not fully visible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Womens satisfaction | 2 hours
  Patients will score their satisfaction by using a 11-step visual analogue scale (VAS) ranging from '0' ("not satisfied at all") to '10' ("very satisfied") 2 hours after Treatment

SECONDARY OUTCOMES:
Postoperative pain | 2 hours
  patients will score their postoperative pain Level using a 11-step visual analogue scale (VAS) ranging from '0' ("no pain" ) to '10' ("maximum pain") within 2 hours after surgery
the resected cone mass | 10 minutes
  the resected cone mass will be quantified by weighing the removed tissue with a precision scale located in the operating room
Operation time | 20 minutes
  the time from the beginning of the Operation (start of the electrosurgical method) until the end of the operation (the end of hemostatic interventions) will be measured in minutes
Operative complications | 14 days
  Operative complications defined as necessity to intervene therapeutically up to 14 days postoperatively
Time to complete intraoperative hemostasis | 120 seconds
  the time until complete hemostasis as judged by the surgeon has been achieved, will be measured in seconds
Surgeons satisfaction | 20 minutes
  Surgeons will score their satisfaction by using a 11-step visual analogue scale (VAS) 20 minutes after Treatment
number of fragments of the surgical specimen | 20 minutes
  surgeons will count the number of the surgical specimen (1 vs. >1)
the dimensions of the surgical specimens | 20 minutes
  The circumference, length and thickness of The surgical specimens will be measured
Intraoperative blood loss | 5 hours
  intraoperative blood loss will be measured using the difference in serum hemoglobin one day prior to surgery and within 5 hours postoperatively
Margin status | 2 days after conization
  Resection margin is judge as "R0" if abnormal cells are not found in the margin of the biopsy or "R1" if abnormal cells remain in the margin of the biopsy. The histopathological examination will be done by an Independent pathologist

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Hilal, M.D., Principal Investigator — Zydolab - Institute of Cytology and Immune Cytochemistry
Locations (1):
- Department of Obstetrics and Gynecology of the Ruhr University Bochum, Herne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rezniczek GA, Hecken JM, Rehman S, Dogan A, Tempfer CB, Hilal Z. Syringe or mask? Loop electrosurgical excision procedure under local or general anesthesia: a randomized trial. Am J Obstet Gynecol. 2020 Dec;223(6):888.e1-888.e9. doi: 10.1016/j.ajog.2020.06.041. Epub 2020 Jul 24. PMID 32585223